CLINICAL TRIAL: NCT04802551
Title: The Effect of Sensory Integration Therapy on Upper Extremity Functions, Trunk Control and Balance in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Hilal AKTAS, Hilal AKTAS, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Izmir Bakircay University
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Sensory integration therapy
- Control group (No Intervention)

INTERVENTIONS:
Other: Sensory integration therapy — Sensory integration disorder is defined as the inability of a person to use the information he / she receives through his / her senses properly in order to continue his daily life properly. Intervention group have some therapy sessions which include sensory integration therapy exercises.
  Arms: Intervention group

SUMMARY:
In children with cerebral palsy, the interactions of the sensory systems, musculoskaletal system and central nervous system are damaged. This situation plays an important role in the realization of trunk control and upper extremity functions.When we look at the literature, it was seen that upper extremity functions were associated with trunk control and oscillation, and it was observed that upper extremity functions were improved in cases with increased trunk control and balance.In the studies, it was concluded that increasing the trunk control improves the static and dynamic balance.Ayres introduced the theory of sensory integrity in the 1970s and defined sensory integration as "the neurological process that organizes the senses coming from the person's body and the environment and makes it possible to use the body effectively in the environment".Sensory integration disorder is defined as the inability of a person to use the information he / she receives through his / her senses properly in order to continue his daily life properly.The incidence of sensory integration disorder in children with motor dysfunction such as cerebral palsy and central nervous system involvement is between 40 and 80%.In children with cerebral palsy, due to central nervous system damage, posture problems, lack of movement and functional deficiencies, sensory problems that can cause balance losses can be seen. When we look at the literature, it has been seen that there are studies on balance, trunk control and upper extremity functions in children with cerebral palsy, but among these studies, the inadequacy of studies that associate balance disorders and trunk control with sensory integration therapy was observed.In this study, the effects of sensory integration therapy on balance, trunk control and upper extremity functions in children with cerebral palsy will be investigated.Pediatric Balance Scale, Trunk Control Measurement Scale, Upper Extremity Skill Quality Scale will be used for balance assessment of individuals with cerebral palsy participating in the study.The study was planned as a single blind randomized control.Participants will be randomly divided into two groups, the control group will be given balance exercises that are included in the standard physiotherapy program, and the experimental group will be given sensory integration exercises for the vestibular system in addition to standard physiotherapy programs.The treatment program to be applied to both experimental and control groups will be carried out by a physiotherapist who has 7 years of experience in pediatric physiotherapy and has 6 years of active sensory integration therapy.Evaluations will be evaluated 3 times by a blinded physiotherapist experienced in the field of pediatrics before, after treatment and 8 weeks after the late period effects.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 0-18
* Being diagnosed with cerebral palsy
* Consent to participate in the study by the parents

Exclusion Criteria:

* Having received botulinum toxin injection in the last 6 months
* Having musculoskaletal surgery in the last 6 months
* Having severe mental retardation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Upper extremity functions | 8 weeks
  It will be measured via Quality of Upper Extremity Skills Test
Trunk Control | 8 weeks
  It will be measured via Trunk Control Measurement Scale
Balance | 8 weeks
  It will be measured via Pediatric Balance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Gulbin ERGIN, Assoc. Prof, Principal Investigator — Izmir Bakircay University
Locations (1):
- Izmir Bakircay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No